CLINICAL TRIAL: NCT01310101
Title: Ofatumumab Added to Dexamethasone in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brno University Hospital (Other)
Collaborators: University Hospital Hradec Kralove (Other); Faculty Hospital Kralovske Vinohrady (Other Government); General Teaching Hospital, Prague (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Michael Doubek, M.D., Ph.D, M.D., Ph.D., Brno University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O-DEX-1, OFA 113815
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Refractory; Relapse; Ofatumumab; Dexamethasone
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — ofatumumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ofatumumab plus dexamethasone (Experimental)
  Interventions: Drug: ofatumumab plus dexamethasone

INTERVENTIONS:
Drug: ofatumumab plus dexamethasone — Dose and schedule
  Cycle 1:
  Ofatumumab: 300 mg as an i.v. infusion on day 1 of the cycle; Ofatumumab: 2000 mg as an i.v. infusion on days 8, 15, 22; Dexamethasone: 40 mg/day p.o., days 1-4 and 15-18
  Cycles 2 to 6 (cycles every 28 days):
  Ofatumumab: 1000 mg i.v. infusion on day 1, 8, 15 and 22 of the cycle; Dexamethasone: 40 mg/day p.o., days 1-4 and 15-18

SUMMARY:
The rationale of the study is to explore the safety and efficacy of ofatumumab in combination with dexamethasone (O-dex regimen) in patients with refractory/relapsed CLL. Moreover, the hypothesis is that this approach will be able to achieve at least the same response rates compared with R-dex regimens (historical controls; manuscript submitted to Leukemia), while maintaining lower toxicity profile.

DETAILED DESCRIPTION:
This is an open-label, multi-center, non-randomized, phase II study to evaluate the safety and efficacy of ofatumumab added to dexamethasone in subjects with relapsed or refractory chronic lymphocytic leukemia.

The treatment will be given for a minimum of 3 cycles, until the best response, or up to a maximum of 6 cycles. After completion of the treatment phase in all patients, survival and disease status assessments will be performed in 1 month post treatment, and then every 2 months for 3 years. The patient will be followed-up in the study for 3 years if there is no progression.

Dose and schedule Cycle 1: Ofatumumab: 300 mg as an i.v. infusion on day 1 of the cycle Ofatumumab: 2000 mg as an i.v. infusion on days 8, 15, 22; Dexamethasone: 40 mg/day p.o., days 1-4 and 15-18; Cycles 2 to 6 (cycles every 28 days): Ofatumumab: 1000 mg i.v. infusion on day 1, 8, 15 and 22 of the cycle; Dexamethasone: 40 mg/day p.o., days 1-4 and 15-18.

Response will be assessed according to the IWCLL guidelines. The investigator assessment of response and progression will be considered primary for all endpoints described in the study.

Safety of the treatment will be evaluated by: adverse events, laboratory tests, vital signs, electrocardiogram and performance status.

Study Endpoints

Primary Endpoint:

Overall response rate (CR, CRi, PR rates)

Secondary Endpoints:

Toxicity, tolerability, adverse events (these events will be assessed by investigator and by the independent reviewers at the key time-points) Overall survival Progression-free survival Time to response and duration of response Time to progression and time to next therapy

Other/Exploratory Endpoints:

Exploratory molecular genetic, immunophenotypic, cytogenetic and pharmacologic markers

ELIGIBILITY:
Inclusion Criteria:

* Male or female previously treated patients with B-cell CLL requiring therapy according to the revised NCI criteria (including CLL patients with immune-mediated hemolysis or thrombocytopenia).
* Flow cytometry confirmation of CLL immunophenotype with CD5, CD19, CD20, CD23, CD79b, and surface Ig at screening.
* Disease recurrence (or refractory disease) after at least one fludarabine-containing regimen, or after at least two previous chemotherapy regimens without fludarabine; and/or poor marrow reserve not allowing chemotherapy administration (Absolute Neutrophil Count < 1.0 x 109/L and/or Absolute Platelet Count < 50 x 109/L).
* Age ≥ 18 years old.
* Signed written informed consent.
* Life expectancy > 3 months.
* ECOG performance status ≤ 2.
* CT scan performed.

Exclusion Criteria:

* Active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study.
* Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
* Prior treatment with anti-CD20 monoclonal antibody or alemtuzumab within 3 months prior to start of therapy.
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C.
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae.
* Known HIV positive.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
* Positive serology for Hepatitis B (HBV) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HBV DNA test will be performed and if positive the subject will be excluded. See section 10.3.2.1 Hepatitis B screening.
* Positive serology for hepatitis C (HCV) defined as a positive test for anti-HCVAb, in which case reflexively perform a HCV RIBA immunoblot assay on the same sample to confirm the result
* Screening laboratory values:

  * creatinine > 2.0 times upper normal limit
  * total bilirubin >1.5 times upper normal limit (unless due to CLL involvement of liver or a known history of Gilbert's disease)
  * ALT > 2.5 times upper normal limit (unless due to disease involvement of liver)
  * alkaline phosphatase > 2.5 times upper normal limit (unless due to disease involvement of the liver or bone marrow)
* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test at screening.
* Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy.
* Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete remission - CR, CRi; partial remission - PR) | Up to Week 24
  The response (CR, CRi, PR rates) will be assessed at the end of therapy of every patient according to international guideline.

SECONDARY OUTCOMES:
Safety profile of the combination of ofatumumab and dexamethasone | Up to Week 24
  Safety of the treatment will be evaluated by: adverse events, laboratory tests, vital signs, electrocardiogram and performance status.
  The safety analysis population will include all subjects who receive at least one dose/infusion and a baseline safety assessment.
Time dependent parameters: progression-free survival (PFS); overall survival (OS). | Year 3 after treatment completion
  PFS and OS will be summarized using Kaplan-Meier plots. Median and the corresponding 95% CI (using Greenwood's formula) will be provided as appropriate. In addition these will be compared with the corresponding plots of a previous study R-dex using one sample log-rank test as described in Finkelstein et al. (J Nat Cancer Inst, 2003).

CONTACTS AND LOCATIONS:
Overall Officials: Jiří Mayer, Prof., M.D., Study Director — University Hospital Brno, Department of Internal Medicine - Hematology and Oncology; Michael Doubek, A.Prof.,M.D., Principal Investigator — University Hospital Brno, Department of Internal Medicine - Hematology and Oncology; Lukáš Smolej, M.D., Ph.D., Principal Investigator — University Hospital Hradec Králové, Department of clinical hematology; Tomáš Kozák, Doc.,M.D., Principal Investigator — University Hospital Královské Vinohrady, Department of clinical hematology; Petra Obrtlíková, M.D., Ph.D., Principal Investigator — Charles University in Prague and General University Hospital in Prague, 1st Department of medicine - Department of hematology
Locations (4):
- Czechia (4):
  - University Hospital Brno, Department of Internal Medicine - Hematology and Oncology, Brno
  - University Hospital Hradec Králové, Department of clinical hematology, Hradec Králové
  - University Hospital Královské Vinohrady, Department of clinical hematology, Prague
  - Charles University in Prague and General University Hospital in Prague, 1st Department of medicine - Department of hematology, Prague

REFERENCES:
- [Derived] Doubek M, Brychtova Y, Panovska A, Sebejova L, Stehlikova O, Chovancova J, Malcikova J, Smardova J, Plevova K, Volfova P, Trbusek M, Mraz M, Bakesova D, Trizuljak J, Hadrabova M, Obrtlikova P, Karban J, Smolej L, Oltova A, Jelinkova E, Pospisilova S, Mayer J. Ofatumumab added to dexamethasone in patients with relapsed or refractory chronic lymphocytic leukemia: Results from a phase II study. Am J Hematol. 2015 May;90(5):417-21. doi: 10.1002/ajh.23964. Epub 2015 Apr 1. PMID 25645263